CLINICAL TRIAL: NCT05565092
Title: A Phase 2a, Randomized, Open-Label Study to Evaluate Multiple Dosing Regimens of Subcutaneous ALXN1820 in Adult Participants With Sickle Cell Disease
Brief Title: Safety, Efficacy, Pharmacokinetic, and Pharmacodynamic Study of ALXN1820 in Adult Participants With Sickle Cell Disease
Acronym: PHOENIX
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision to terminate program.
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ALXN1820-SCD-201; 2022-001615-74 (EudraCT Number)
Record Dates: First submitted 2022-09-15; First posted 2022-10-04 (Actual); Results first posted 2025-01-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Sickle Cell Disease (SCD)
Keywords: Sickle Cell Disease; ALXN1820; SCD
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- ALXN1820 300 mg once weekly (Experimental): Participants will receive 300 milligrams (mg) once weekly (QW).
  Interventions: Drug: ALXN1820
- ALXN1820 600 mg once every 4 weeks (Experimental): Participants will receive 600 mg once every 4 weeks (Q4W).
  Interventions: Drug: ALXN1820
- ALXN1820 300 mg once every 2 weeks (Optional cohort) (Experimental): Participants will receive 300 mg once every 2 weeks (Q2W).
  Interventions: Drug: ALXN1820

INTERVENTIONS:
Drug: ALXN1820 — ALXN1820 will be administered subcutaneously.

SUMMARY:
The primary objective of this study is to assess the safety and tolerability of ALXN1820 SC (subcutaneous) in participants with SCD (Sickle Cell Disease).

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of SCD (HbSS, or HbSβ0-thalassemia).
* Body weight ≥ 40 kg (inclusive) at Screening.
* Must follow protocol-specified contraception guidance while on treatment and for up to 6 months after last dose.
* Hemoglobin between 5.5 and 10 g/dL at Screening
* Have had 1 to 10 VOCs in the past 12 months.
* Patients receiving hydroxyurea must have been on a stable dose for ≥ 3 months prior to providing informed consent, with no anticipated need for dose adjustment during the study.
* Patients will be vaccinated with MCV4 and serogroup B meningococcal vaccinations at least 14 days before dosing, if not already vaccinated within 3 years before the first dose.
* Haemophilus influenzae type b (Hib) and Streptococcus pneumoniae vaccination are up to date according to current national/local vaccination guidelines for patients with SCD.

Exclusion Criteria:

* Planned initiation, termination, or dose alteration of hydroxyurea during the study.
* Receiving Voxelotor (OXBRYTA) or crizanlizumab (ADAKVEO) within 60 days of providing informed consent.
* Receiving treatment with recombinant human erythropoetins (eg, epoetin alfa).
* Treated with complement inhibitors within 6 months prior to the first dose.
* Patients who are on chronic transfusion or receive a transfusion within 60 days of first dose.
* Any significant disease or disorder which, in the opinion of the Investigator, may put the participant at risk.
* Hepatitis B (positive hepatitis surface antigen [HBsAg] or positive core antibody (anti-HBc) with negative surface antibody [anti-HBs]) or hepatitis C viral infection (hepatitis C virus [HCV] antibody positive, except for patients with documented successful treatment and documented sustained virologic response) at Screening.
* Active systemic bacterial, viral, or fungal infection within 14 days prior to dosing.
* Participation (ie, last protocol-required study visit) in a clinical study within 90 days or 5 half-lives of the investigational agent, whichever is longer, before initiation of dosing on Day 1.
* Participation in more than 1 clinical study of a monoclonal antibody (mAb), or participation in a clinical study of a mAb within the 6 months or 5 half-lives of the mAb, whichever is longer, prior to Screening, during which the participant was exposed to the active study drug.
* Severe renal impairment (estimated glomerular filtration rate [eGFR] < 30 mL/min/1.73 m2 ) or on chronic dialysis.
* History of allergy or hypersensitivity to excipients of ALXN1820 (eg, polysorbate 80).
* History of complement deficiency.
* History of N meningitidis, S pneumoniae, or H influenzae infection.
* History of malignancy with the exception of a nonmelanoma skin cancer or carcinoma in situ of the cervix that has been treated with no evidence of recurrence within 5 years.
* Participants who are pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2023-02-22 (Actual); Primary Completion 2024-01-09 (Actual); Study Completion 2024-01-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Research Site, Hollywood, Florida
  - Research Site, Indianapolis, Indiana

IPD SHARING:
Plan to Share IPD: Yes
Alexion has a public commitment to allow requests for access to study data and will be supplying a protocol, CSR, and plain language summaries.
Supporting Information: Study Protocol, SAP, CSR

REFERENCES:
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=ALXN1820-SCD-201&attachmentIdentifier=7594508e-5c80-45fc-8d21-19e19a57ef58&fileName=alxn1820-scd-201-Protocol_amendment_1.0_redacted_14Aug2023.pdf&versionIdentifier=
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=ALXN1820-SCD-201&attachmentIdentifier=233055bd-e074-4215-8b2f-1575d7291e2a&fileName=ALXN1820-SCD-201_SAP_V1.0_24Oct2023_final_redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Per Sponsor decision, the study was terminated. Only 2 participants were enrolled. Due to concerns regarding participant confidentiality, no data are reported.
Groups:
- ALXN1820 300 mg QW: Participants received 300 milligrams (mg) once weekly (QW).
- ALXN1820 600 mg Q4W: Participants received 600 mg once every 4 weeks (Q4W).
- ALXN1820 300 mg Q2W (Optional Cohort): Participants received 300 mg once every 2 weeks (Q2W).
Period: Overall Study
Arm/Group | ALXN1820 300 mg QW | ALXN1820 600 mg Q4W | ALXN1820 300 mg Q2W (Optional Cohort)
Started | 0 | 0 | 0
Completed | 0 | 0 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Per Sponsor decision, the study was terminated. Only 2 participants were enrolled. Due to concerns regarding participant confidentiality, no data are reported.
Groups:
- ALXN1820 300 mg QW: Participants received 300 mg QW.
- ALXN1820 600 mg Q4W: Participants received 600 mg Q4W.
- ALXN1820 300 mg Q2W (Optional Cohort): Participants received 300 mg Q2W.
- Total: Total of all reporting groups
Arm/Group | ALXN1820 300 mg QW | ALXN1820 600 mg Q4W | ALXN1820 300 mg Q2W (Optional Cohort) | Total
Number analyzed (Participants) | 0 | 0 | 0 | 0
Age, Categorical
Sex: Female, Male
Ethnicity (NIH/OMB)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events and Serious Adverse Events
Time Frame: Baseline through Day 211 (Cohorts 1 and 2) and through Day 169 (Optional Cohort 3)
Population: as for baseline characteristics
Arm/Group | ALXN1820 300 mg QW | ALXN1820 600 mg Q4W | ALXN1820 300 mg Q2W (Optional Cohort)
Number analyzed (Participants) | 0 | 0 | 0

2. Secondary Outcome: Pharmacokinetics: Serum ALXN1820 Concentration
Time Frame: Baseline through Day 211 (Cohorts 1 and 2) and through Day 169 (Optional Cohort 3)
Population: as for baseline characteristics
Arm/Group | ALXN1820 300 mg QW | ALXN1820 600 mg Q4W | ALXN1820 300 mg Q2W (Optional Cohort)
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Change From Baseline in Serum Concentration of Total and Free Properdin Through Day 211 (Cohorts 1 and 2) and Day 169 (Optional Cohort 3)
Time Frame: Baseline through Day 211 (Cohorts 1 and 2) and Day 169 (Optional Cohort 3)
Population: as for baseline characteristics
Arm/Group | ALXN1820 300 mg QW | ALXN1820 600 mg Q4W | ALXN1820 300 mg Q2W (Optional Cohort)
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Change From Baseline Complement Alternative Pathway Activity Through Day 211 (Cohorts 1 and 2) and Day 169 (Optional Cohort 3)
Time Frame: Baseline through Day 211 (Cohorts 1 and 2) and Day 169 (Optional Cohort 3)
Population: as for baseline characteristics
Arm/Group | ALXN1820 300 mg QW | ALXN1820 600 mg Q4W | ALXN1820 300 mg Q2W (Optional Cohort)
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: Change From Baseline in Complement Biomarkers Through Week 12 (Cohorts 1 and 2)
Time Frame: Baseline, Week 12
Population: as for baseline characteristics
Arm/Group | ALXN1820 300 mg QW | ALXN1820 600 mg Q4W | ALXN1820 300 mg Q2W (Optional Cohort)
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Change From Baseline in Hemoglobin Level at Week 12 (Cohorts 1 and 2)
Time Frame: Baseline, Week 12
Population: as for baseline characteristics
Arm/Group | ALXN1820 300 mg QW | ALXN1820 600 mg Q4W | ALXN1820 300 mg Q2W (Optional Cohort)
Number analyzed (Participants) | 0 | 0 | 0

7. Secondary Outcome: Change From Baseline in Hemolysis Markers at Week 12 (Cohorts 1 and 2)
Time Frame: Baseline, Week 12
Population: as for baseline characteristics
Arm/Group | ALXN1820 300 mg QW | ALXN1820 600 mg Q4W | ALXN1820 300 mg Q2W (Optional Cohort)
Number analyzed (Participants) | 0 | 0 | 0

8. Secondary Outcome: Change From Baseline in Hemopexin at Week 12 (Cohorts 1 and 2)
Time Frame: Baseline, Week 12
Population: as for baseline characteristics
Arm/Group | ALXN1820 300 mg QW | ALXN1820 600 mg Q4W | ALXN1820 300 mg Q2W (Optional Cohort)
Number analyzed (Participants) | 0 | 0 | 0

9. Secondary Outcome: Number of Participants With Antidrug Antibodies to ALXN1820
Time Frame: Baseline through Day 211 (Cohorts 1 and 2) and through Day 169 (Optional Cohort 3)
Population: as for baseline characteristics
Arm/Group | ALXN1820 300 mg QW | ALXN1820 600 mg Q4W | ALXN1820 300 mg Q2W (Optional Cohort)
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Per Sponsor decision, the study was terminated. Only 2 participants were enrolled. Due to concerns regarding participant confidentiality, no data are reported.
Description: Per Sponsor decision, the study was terminated. Only 2 participants were enrolled. Due to concerns regarding participant confidentiality, no data are reported.
Arm/Group | ALXN1820 300 mg QW | ALXN1820 600 mg Q4W | ALXN1820 300 mg Q2W (Optional Cohort)
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Per Sponsor decision, the study was terminated. Only 2 participants were enrolled. Due to concerns regarding participant confidentiality, no data are reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-08-14): https://cdn.clinicaltrials.gov/large-docs/92/NCT05565092/Prot_002.pdf
  • Statistical Analysis Plan (2023-10-24): https://cdn.clinicaltrials.gov/large-docs/92/NCT05565092/SAP_001.pdf